CLINICAL TRIAL: NCT00006254
Title: A Phase I Trial of a Live, Genetically Modified Salmonella Typhimurium (VNP20009) for the Treatment of Cancer by Intravenous Administration
Brief Title: VNP20009 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-008; CDR0000068187 (Registry Identifier: PDQ (Physician Data Query)); CCF-IRB-3663; NCI-V00-1622
Record Dates: First submitted 2000-09-11; First posted 2003-09-03 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2007-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — VNP 20009

INTERVENTIONS:
Biological: salmonella VNP20009

SUMMARY:
RATIONALE: Biological therapies such as VNP20009 use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I trial to study the effectiveness of VNP20009 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose or minimum effective dose and associated toxic effects of VNP20009 in patients with advanced solid tumors.
* Determine whether VNP20009 can be detected in tumors after treatment in these patients.
* Determine the pharmacokinetics of this treatment regimen in these patients.
* Determine the antitumor effects of this treatment regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive VNP20009 IV over 4 hours on day 1. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable disease or partial or complete response (CR) may receive additional courses every 35 days for up to 12 total doses or 2 courses past a CR.

Cohorts of 3-6 patients receive escalating doses of VNP20009 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6-9 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 14-45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced and/or metastatic solid tumors refractory to standard curative or palliative therapy and for which no other conventional therapy exists
* Measurable or evaluable metastatic disease
* No brain metastases unless previously treated and no evidence of recurrence
* No lymphoma or other hematologic malignancy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hematocrit at least 30% (transfusion allowed)
* No known bleeding disorder

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 1.5 times ULN (3 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 1.5 times ULN (3 times ULN if liver metastases present)
* PT and PTT no greater than 1.5 times ULN
* Hepatitis B surface antigen negative
* No chronic active hepatitis B
* No end-stage liver disease

Renal:

* Creatinine no greater than 2.0 mg/dL
* No urinary tract stones
* No end-stage renal disease

Cardiovascular:

* No known valvular disease
* No known clinically significant atherosclerotic disease, peripheral vascular disease, or arterial aneurysm
* No unstable angina
* No artificial heart valves

Pulmonary:

* No severe oxygen-dependent chronic obstructive pulmonary disease

Other:

* No artificial implant that cannot be removed (e.g., prosthetic hips or knees or other devices)
* No permanent central venous catheters
* No gallstones
* No active infection
* No documented Salmonella infection
* No tumor fever or fever of unknown origin or cause
* Daily maximum temperature no greater than 38.0 degrees Celsius
* HIV negative
* No documented immunodeficiency
* No other life-threatening illness
* No history of allergic reaction or hypersensitivity to quinolone or cephalosporin antibiotics
* No commercial food handlers, day-care workers, or health-care workers
* No patients unable to avoid close personal contact with severely immunosuppressed individuals (e.g., other patients on myelosuppressive cancer chemotherapy)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered

Chemotherapy:

* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered

Endocrine therapy:

* At least 2 weeks since prior hormonal therapy and recovered
* No concurrent steroids that could depress the immune system unless indicated for severe reactions

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* At least 2 weeks since prior surgery and recovered
* No prior splenectomy
* No concurrent palliative surgery

Other:

* Recovered from any other prior anticancer therapies
* No concurrent antibiotics
* No concurrent immunosuppressives or any other medications that could suppress the immune system
* No other concurrent treatment for malignancy
* No requirement for immediate palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio